CLINICAL TRIAL: NCT05919719
Title: Fluid Responsiveness Evaluation by a Non-invasive Method in CHildren - The FRENCH Study
Brief Title: Fluid Responsiveness Evaluation by a Non-invasive Method in CHildren
Acronym: FRENCH
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/48
Record Dates: First submitted 2023-06-02; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Circulatory Failure (Shock)
Keywords: shock; volume expansion; goal-directed fluid management; echocardiography
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study of diagnostic accuracy: Patients included in this study would have received fluid expansion in all cases, as the prescription of 10 to 20ml/kg crystalloid fluid expansion by the physician in charge is the main inclusion criterion.
  Interventions: Procedure: Non interventional study (study of diagnostic accuracy with an extra echocardiographic assessment).

INTERVENTIONS:
Procedure: Non interventional study (study of diagnostic accuracy with an extra echocardiographic assessment). — Fluid expansion will be delayed while our index test is performed. After fluid expansion, patient will undergo an echocardiographic assessment of response to fluid expansion (gold-standard).
  Our index test is the ΔSVi-AC: indexed percentage of stroke volume variation between baseline and during a standardized abdominal compression. Stroke volume will be assessed by transthoracic echocardiography.
  Patient will undergo 3 echocardiographic assessment: At baseline, During abdominal compression, After the 10 to 20ml/kg crystalloid fluid expansion Abdominal compression : a sphygmomanometer will be inflated to a pressure of less than 10 mmHg and will be applied to the center of the patient's abdomen. Then, a gentle compression on the sphygmomanometer will be performed, calibrated at 22 - 26 mmHg according to the sphygmomanometer. The echocardiographic assessments will take place between 10 and 60 seconds after the start of the compression, which will therefore last less than a minute.

SUMMARY:
In this study, the investigators aim to validate a non-invasive marker of fluid-responsiveness in children with acute circulatory failure based on standardized abdominal compression. This would allow physicians to identify which patient could benefit from a fluid expansion, thus avoiding a potentially useless or even dangerous fluid expansion, leading to fluid overload. To this end, the investigators will evaluate the diagnostic accuracy (sensitivity and specificity) of stroke volume variation induced by standardized abdominal compression for the diagnosis of fluid responsiveness (based on the gold-standard test: significant increase in cardiac index after fluid expansion).

DETAILED DESCRIPTION:
Fluid expansion is the cornerstone of acute circulatory failure treatment in children Although this therapy drastically reduced mortality, several studies in recent years have highlighted the adverse effects of excessive fluid expansion (leading to fluid overload). Currently, the search for indicators to predict fluid responsiveness is a major issue in intensive care. These indicators are based on Franck-Starling's law: if small changes in preload lead to an increase in cardiac output, then fluid responsiveness can be expected. However, in children, the only validated indicator (respiratory variability of peak aortic velocity) can only be used in the absence of any spontaneous respiratory movement, a rare situation in practice. Recently, two pediatric studies investigated a simple clinical test: hepatic or abdominal compression. This clinical maneuver, by increasing venous return via mobilization of the hepato-splanchnic reserve, induces a transient and reversible preload increase. The evaluation of the hemodynamic effects of this "endogenous fluid expansion" allowed, according to the authors, to accurately predict fluid responsiveness. However, several factors reduce the applicability of these results: the small number of studies on this subject, the smaller volume of fluid used than in clinical practice, and the population studied, composed almost exclusively of children in postoperative of cardiac surgery.

In this study, the investigators will evaluate the diagnostic accuracy of abdominal compression for the diagnosis of fluid responsiveness in children with acute circulatory failure, hospitalized in pediatric intensive care unit (PICU) for a medical or a non-cardiac surgical condition, for whom a fluid expansion was prescribed by the physician in charge. The index test will be the stroke volume variation following a standardized abdominal compression (before fluid expansion). The gold standard test will be the variation of cardiac output between baseline and after fluid expansion, a variation > 15% defining fluid responsiveness.

In this non interventional study of diagnostic accuracy, patients will undergo an extra echocardiographic assessment, but no supplemental blood test or invasive parameters will be collected. Simple clinical parameters will be collected within 4 hours after the fluid expansion. Patients will be follow-up until PICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age lower than 15 years old
* Prescription of a 10 to 20ml/kg crystalloid fluid expansion by the physician in charge
* Acute circulatory failure defined by the association of an A criteria (increase of heart rate more than two standard deviation for the age, decrease of systolic or mean blood pressure more than two standard deviation for ) and a B criteria (lactate more than 2 mmol/L, oliguria less than 1mL/kg/h, a capillary filling time more than 3 seconds, mottling)
* Patient hospitalized in PICU

Exclusion Criteria:

* Prematurity (term below 37 gestational week).
* Acute cardiogenic pulmonary edema
* Hemodynamic instability making the delay necessary for abdominal compression and ultrasonography dangerous for the patient
* Non corrected congenital cardiopathy, or inferior to 15 days postoperative.
* Intra-abdominal hypertension or painful abdominal palpation
* Abdominal surgery in the last 15 days
* Supine position contraindicated or deleterious
* No investigator available to assess ultrasonographic measures
* Impairment of echocardiographic acoustic window or restless patient making ultrasonography impossible

Ages: 1 Minute to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: At least 24 fluid expansion are needed, in 10 to 24 patients (maximum of 3 fluid expansion per patient). The "number needed to treat" was calculated with Obuchowski method, with an aphla risk of 0.05, a statistical power of 80%, a ratio "responder/nonresponder" of 1:1, and a predicted area under the receiver operating characteristic curve of 0.78 (based on previous studies).
  In order to be clinically relevant, since a large majority of patients admitted to our PICU are under 2 years of age, the investigators plan to include 24 fluid expansions administrated to patients under 2 years old. Therefore, the investigators might include more than 24 fluid expansions if some are administrated to patients older than 2 years old. Without this correction, our study might be underpowered if age is found to be a bias in fluid responsiveness.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the index test (ΔSVi-AC) for the diagnosis of fluid responsiveness | after abdominal compression, 30 minutes to 4 hours after baseline
  Diagnostic accuracy of the index test (ΔSVi-AC) for the diagnosis of fluid responsiveness, defined by an increase of cardiac output > 15% after fluid expansion (ΔCO-FE > 15%, gold-standard test) Index test (ΔSVi-AC) will be calculated as the difference between Stroke Volume (SV) after abdominal compression and SV at baseline, divided by SV at baseline (%). SV will be measured by echocardiographic assessment.
  Gold-standard test (ΔCO-FE) will be calculated as the difference between CO after fluid expansion and CO at baseline, divided by CO at baseline (%). CO will be measured by echocardiographic assessment.

SECONDARY OUTCOMES:
Association between elevated ΔSVi-AC and capillary filling time (sec) -Baseline | at baseline (before fluid expansion)
  Association between elevated ΔSVi-AC and capillary filling time (sec). Normal value: < 3 seconds
Association between elevated ΔSVi-AC and capillary filling time (sec) -after abdominal compression | after abdominal compression, 30 minutes to 4 hours after baseline
  Association between elevated ΔSVi-AC and capillary filling time (sec). Normal value: < 3 seconds.
Association between elevated ΔSVi-AC and Heart rate (bpm). -Baseline | at baseline (before fluid expansion)
  Association between elevated ΔSVi-AC and Heart rate (bpm). Normal value: < 2 standard deviation for the age
Association between elevated ΔSVi-AC and Heart rate (bpm). -after abdominal compression | after abdominal compression, 30 minutes to 4 hours after baseline
  Association between elevated ΔSVi-AC and Heart rate (bpm). Normal value: < 2 standard deviation for the age
Association between elevated ΔSVi-AC and Mean blood pressure (mmHg). -Baseline | at baseline (before fluid expansion)
  Association between elevated ΔSVi-AC and Mean blood pressure (mmHg). Normal value: < 2 standard deviation for the age
Association between elevated ΔSVi-AC and Mean blood pressure (mmHg). -after abdominal compression | after abdominal compression, 30 minutes to 4 hours after baseline
  Association between elevated ΔSVi-AC and Mean blood pressure (mmHg). Normal value: < 2 standard deviation for the age
Association between elevated ΔSVi-AC and urine output (ml/kg/h). -Baseline | at baseline (before fluid expansion)
  Association between elevated ΔSVi-AC and Urine output (ml/kg/h). Normal value: > 1ml/kg/h.
Association between elevated ΔSVi-AC and urine output (ml/kg/h). -after abdominal compression | after abdominal compression, 30 minutes to 4 hours after baseline
  Association between elevated ΔSVi-AC and Urine output (ml/kg/h). Normal value: > 1ml/kg/h.
Association between elevated ΔSVi-AC and Blood lactate (mmol/L). -Baseline | at baseline (before fluid expansion)
  Association between elevated ΔSVi-AC and Blood lactate (mmol/L). Normal value: < 2mmol/L
Association between elevated ΔSVi-AC and Blood lactate (mmol/L). -after abdominal compression | after abdominal compression, 30 minutes to 4 hours after baseline
  Association between elevated ΔSVi-AC and Blood lactate (mmol/L). Normal value: < 2mmol/L
Association between elevated ΔSVi-AC and Central venous oxygen saturation (%). -Baseline | at baseline (before fluid expansion)
  Association between elevated ΔSVi-AC and Central venous oxygen saturation (%). Normal value: >70%
Association between elevated ΔSVi-AC and Central venous oxygen saturation (%). -after abdominal compression | after abdominal compression, 30 minutes to 4 hours after baseline
  Association between elevated ΔSVi-AC and Central venous oxygen saturation (%). Normal value: >70%

CONTACTS AND LOCATIONS:
Overall Officials: Julien GOTCHAC, MD, Principal Investigator — Bordeaux hospital University
Locations (1):
- Bordeaux Hospital University, Bordeaux, France

REFERENCES:
- [Derived] Gotchac J, Navion A, Belaroussi Y, Klifa R, Amedro P, Guichoux J, Brissaud O. Clinical value of calibrated abdominal compression plus transthoracic echocardiography to predict fluid responsiveness in critically ill infants: a diagnostic accuracy study. BMC Pediatr. 2025 May 7;25(1):361. doi: 10.1186/s12887-025-05728-z. PMID 40329198